CLINICAL TRIAL: NCT00137930
Title: Compare the Immunogenicity, Reactogenicity & Safety of 2 Different Formulations of GSK Biologicals' Live Attenuated Human Rotavirus (HRV) Vaccine Given as a Two-dose Primary Vaccination in Healthy Infants Previously Uninfected With HRV
Brief Title: Study of Immunogenicity & Safety of 2 Different Formulations of Human Rotavirus (HRV) Vaccine for the Prophylaxis of Rotavirus Gastroenteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 104480
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
Keywords: Prophylaxis of rotavirus gastroenteritis
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: Live attenuated rotavirus vaccine

SUMMARY:
Rotavirus (RV) is the most important cause of acute gastroenteritis (GE) requiring the hospitalization of infants and young children in developed and developing countries and can be a frequent cause of death in children less than 5 years of age (estimated nearly 500,000 annual deaths worldwide). GlaxoSmithKline (GSK) Biologicals has developed a vaccine against human rotavirus gastroenteritis. A new formulation of the vaccine, with an alternative buffer, was developed. This study will be conducted to evaluate the new formulation compared to the existing formulation of the HRV vaccine.

DETAILED DESCRIPTION:
The study consists of four groups of children recruited in different centers in Finland. One group of children will receive the existing formulation of HRV vaccine and one group will receive the new formulation of the HRV vaccine. The other two groups will receive the placebo for existing formulation or the new formulation based on the allocation. The vaccine or placebo will be administered starting at 6 - 12 weeks of age according to 0, 1 month schedule. Routine childhood vaccinations are allowed according to local practice, but at least 14 days apart from each dose of study vaccine. The duration of the study will be approximately 2 months per child.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with parents/guardians who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* Males or females between, and including, 6 and 12 weeks (42 - 90 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parents or guardians of the subjects.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration of a vaccine (including routine paediatric vaccines) not foreseen by the study protocol during the period starting from 14 days before each dose of study vaccine(s) and ending 14 days after.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device)
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth. (For corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract or other serious medical condition, as determined by the investigator.
* History of allergic diseases or reactions likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required).
* Major congenital defects or serious chronic illnesses.
* Acute disease at time of enrolment. (Acute disease is defined as the presence of moderate or severe illness with or without fever, i.e. temperature >= 37.5°C as measured by an axillary thermometer or >= 38.0°C as measured by a rectal thermometer.) Temperature greater than or equal to these cut-offs warrants deferral of the vaccination pending recovery of the subject.
* Gastroenteritis (GE) within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Household contact with an immunosuppressed individual or pregnant woman.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.
* Previous confirmed occurrence of RV GE.
* History of neurological disorders or seizures.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250
Dates: Start 2005-08; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Endpoint: immunogenicity and reactogenicity
Proportion of subjects with vaccine take

SECONDARY OUTCOMES:
Proportion of seroconverters
RV-IgA concentration
Occurrence of solicited symptoms: loss of appetite, fussiness/irritability, fever, diarrhea, vomiting, cough/runny nose
Unsolicited symptoms and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Finland (5):
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Debrus S et al. Study of the viral activity of RIX4414 - human rotavirus vaccine. Abstract presented at the 47th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC). Chicago, USA, 17-20 September 2007.
- [Background] Debrus S et al. Viral shedding (methodology). Abstract presented at the 47th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC). Chicago, USA, 17-20 September 2007.
- [Background] Vesikari T et al. Immunogenicity of liquid formulation of the oral live attenuated human rotavirus vaccine (Rotarix™). Abstract presented at the 12th Annual Congress of Sociedad Latinoamericana de Infectología Pediátrica (SLIPE). San Jose, Costa Rica 8-11 May 2007.
- [Derived] Vesikari T, Karvonen A, Bouckenooghe A, Suryakiran PV, Smolenov I, Han HH. Immunogenicity, reactogenicity and safety of the human rotavirus vaccine RIX4414 oral suspension (liquid formulation) in Finnish infants. Vaccine. 2011 Mar 3;29(11):2079-84. doi: 10.1016/j.vaccine.2011.01.004. Epub 2011 Jan 14. PMID 21238572
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register